CLINICAL TRIAL: NCT06518070
Title: Results Comparison of Cervical Cancer Early Detection Using Cerviray With VIA Test
Status: Completed | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Other Study IDs: OBGY-202405.01
Record Dates: First submitted 2024-06-01; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; cerviray; via test; early detection
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cerviray AI — Patient was screened using Cerviray AI, Cerviray AI evaluation by expert anc compared to VIA test in the same day.

SUMMARY:
Cervical cancer, primarily caused by Human Papilloma Virus (HPV), is a significant global health concern, ranking as the fourth most common cancer in women worldwide. In Indonesia, it stands as the second most frequent cancer among women. This study investigates the performance of Cerviray® AI and Cerviray® AI Evaluation, an artificial intelligence (AI) technology for diagnosing cervical cancer, aiming to compare its sensitivity, specificity, positive predictive value (PPV), and area under the receiver operating characteristic curve (AUC ROC) with the Visual Inspection with Acetic Acid (VIA) test.

DETAILED DESCRIPTION:
The study involved 44 patients from various health centers in West Java Province. Cerviray® AI, Cerviray® AI Evaluation, and VIA tests were administered to high-risk women of childbearing age.

ELIGIBILITY:
Inclusion Criteria:

* high-risk women of childbearing age who would be screened for cervical cancer (by Cerviray AI examination, Cerviray AI evaluation, and VIA test) at 1 clinic and other 4 health centers

Exclusion Criteria:

* incomplete data
* patient refusing to be examined
* patient refusing to participate in the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cancer cervix is only limited in female patient
Study Population: women of childbearing age who would be screened for cervical cancer in West Java Province
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Cerviray AI | 1 day
  The target population screened using Cerviray AI tools and Cerviray AI evaluation and will be compared to VIA test and confirmed by the anatomical pathology examination. The data will be shown as analytical results of the Cerviray AI tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Padjajaran University, Bandung, Indonesia

REFERENCES:
- [Derived] Harsono AB, Susiarno H, Suardi D, Mantilidewi KI, Wibowo VD, Hidayat YM. Results comparison of cervical cancer early detection using cerviray (R) with VIA test. BMC Res Notes. 2025 Jan 22;18(1):30. doi: 10.1186/s13104-025-07086-6. PMID 39844244